CLINICAL TRIAL: NCT04172246
Title: A Phase 1/2 Study of Zanubrutinib in Japanese Patients With Mature B-Cell Malignancies
Brief Title: Study of Zanubrutinib in Japanese Participants With B-Cell Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-111; JapicCTI-195047 (Registry Identifier: Jape)
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Mature B-cell Malignancies
Keywords: relapsed/refractory chronic lymphocytic leukemia; relapsed/refractory small lymphocytic lymphoma; treatment-naïve chronic lymphocytic leukemia; treatment-naïve /small lymphocytic lymphoma; relapsed/refractory mantle cell lymphoma; relapsed/refractory marginal zone lymphoma; relapsed/refractory follicular lymphoma; relapsed/refractory Waldenström macroglobulinemia; treatment-naïve Waldenström macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental)
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib at 160 mg orally twice daily
  Other Names: BGB-3111

SUMMARY:
This is a Phase 1/2 study of zanubrutinib in Japanese participants with mature B-cell malignancies.

This study intends to assess the use of zanubrutinib as an investigational agent to develop new treatment options for Japanese participants with B-cell malignancies. No formal hypothesis testing will be performed given the small sample size.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with Confirmed diagnosis of mature B-cell neoplasms including chronic lymphocytic leukemia/ small lymphocytic lymphoma, mantle cell lymphoma, follicular lymphoma, marginal zone lymphoma and Waldenström's macroglobulinemia
* Relapsed/refractory disease defined as disease that relapsed after, or been refractory to, at least 1 prior therapy
* Meeting at least one of criteria for requiring treatment
* Measurable disease by computed tomography (CT)/ magnetic resonance imaging (MRI) for mantle cell lymphoma (MCL), marginal zone lymphoma (MZL) and follicular lymphoma (FL) participants and by serum immunoglobulin (Ig) M level > 0.5 g/dL for WM participants
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Life expectancy of > 4 months

Key Exclusion Criteria:

* Known central nervous system involvement by lymphoma/leukemia
* Known plasma cell neoplasm, prolymphocytic leukemia, history of or currently suspected Richter's syndrome
* Prior allogeneic stem cell transplant
* Systemic chemotherapy or radiation therapy within 2 weeks prior to first dose of zanubrutinib
* Active fungal, bacterial, and/or viral infection requiring systemic therapy
* Prior therapy with B-cell receptor inhibitor (eg, Bruton tyrosine kinase, phosphoinositide 3 kinase delta, and/or spleen tyrosine kinase inhibitor) or B-cell lymphoma 2 inhibitor (eg, venetoclax/ABT-199)
* Pregnant, lactating, or nursing women
* Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 1: Number of Participants Experiencing Treatment-Emergent Serious Adverse Events (SAEs) | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 1: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation of Treatment | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 1: Maximum Plasma Concentration (Cmax) of zanubrutinib | Up to 29 days
Part 1: Area under plasma concentration-time curve Concentration (AUC) of zanubrutinib | Up to 29 days
Part 2: Overall response rate as assessed by Independent Review Committee (IRC) | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever occurs first

SECONDARY OUTCOMES:
Part 1: Bruton tyrosine kinase (BTK) occupancy in peripheral blood mononuclear cells | Predose up to 24 hours postdose
Part 1: Overall response rate (ORR) as assessed by the investigator | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 1: Progression-free survival (PFS) as assessed by the investigator | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 1: Duration of response as assessed by the investigator | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 1: Time to response as assessed by the investigator | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Number of Participants Experiencing Treatment-Emergent Serious Adverse Events (SAEs) | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Maximum Plasma Concentration (Cmax) of zanubrutinib | Predose up to 24 hours postdose Cycle 1 day 1 (C1D1) and Cycle 2 day 1 (C2D1)
Part 2: Number of Participants Experiencing AEs Leading to Discontinuation of Treatment | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Rate of complete response for chronic lymphocytic leukemia (CLL) as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Rate of complete response with incomplete marrow for CLL as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Rate of complete response for small lymphocytic lymphoma (SLL), mantle cell lymphoma (MCL), and Waldenström macroglobulinemia (WM) as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Rate of very good partial response (VGPR) or better for WM as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Major response rate (partial response or better) for WM as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Rate of partial response or better for CLL as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Overall response rate (ORR) by disease type as assessed by the investigator | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Progression-free survival (PFS) as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Duration of response as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
Part 2: Time to response as assessed by IRC | Until approximately 6 months after the last dose of zanubrutinib for the last participant who discontinues zanubrutinib or zanubrutinib becomes commercially available for the participant's disease, whichever is earlier
To assess the efficacy of zanubrutinib as measured by overall survival | Overall survival defined as time from start of study treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (15):
- Japan (15):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashishi, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Kurume University Hospital, KurumeShi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Aiiku Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, KobeShi, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Cancer Center Hospital, ChuoKu, Tokyo
  - Aomori Prefectural Central Hospital, Aomori
  - Gifu Municipal Hospital, Gifu
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - National Hospital Organization Okayama Medical Center, Okayama
  - Yokohama Municipal Citizens Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/